CLINICAL TRIAL: NCT03699631
Title: PROACTIVE: Prevention of Acute and Chronic GVHD Using TocIlizumab in Combination With Standard GVHD Prophylaxis After allogEneic Transplantation
Brief Title: PROACTIVE: Preventing Acute/Chronic GVHD With TocIlizumab Combined With GVHD Prophylaxis Post allogEneic Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William R. Drobyski, MD, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO32694; 1K08HL143189-01A1 (NIH); 5P30CA008748 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Tacrolimus; Methotrexate; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tacrolimus/Methotrexate/Tocilizumab (Experimental): Patients enrolled on the clinical trial will receive tacrolimus initiating at Day -1 at doses to maintain therapeutic levels per institutional preference and continued until at least Day +90 post-transplant.
  Methotrexate will be administered intravenously and dosed at 15 mg/m2 Day +1 and 10 mg/m2 Days +3, +6 and +11.
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg on Day -1 and at day +100 (+/- 14 days).
  Interventions: Drug: Tacrolimus; Drug: Methotrexate; Drug: Tocilizumab

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus will be given intravenously at a dose of 0.03 mg/kg/day starting Day -3. Subsequent dosing will be based on blood levels.
  Other Names: Prograf
Drug: Methotrexate — Methotrexate will be administered at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic cell infusion.
  Other Names: Trexall
Drug: Tocilizumab — Tocilizumab will be administered intravenously (IV) at a dose of 8 mg/kg (maximum dose of 800 mg) once on the Day -1 approximately 24 hours prior to the estimated time of the hematopoietic cell infusion, and subsequently, on Day +100 (+/- 14 days, i.e., Days +86 to +114) post-alloHCT. The infusion will be administered over 60 minutes through a dedicated IV line and must not be administered by IV bolus.
  Other Names: Actemra

SUMMARY:
This is a phase II open-label trial designed to evaluate the efficacy of tocilizumab in improving GVHD-free/relapse-free survival (GRFS) after allogeneic hematopoietic cell transplantation (alloHCT) for hematologic malignancy.

DETAILED DESCRIPTION:
The research team earlier hypothesized and demonstrated that tocilizumab could attenuate the incidence of acute GVHD (aGVHD) after myeloablative conditioning (MAC) and reduced intensity conditioning (RIC) Allogeneic hematopoietic cell transplantation (alloHCT), using matched sibling or unrelated donor. In this study, the research team hypothesizes that longer term interleukin 6 (IL-6) inhibition through treatment with tocilizumab by repeated dosing would mediate a beneficial effect not only on the risk of aGVHD, but also on chronic GVHD. This will be achieved by administering an additional dose of tocilizumab at Day +100 post-alloHCT, besides the pretransplant dose, as done in our previous clinical trial, thereby providing total prophylaxis against both acute and chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients with any hematologic malignancy for which alloHCT is indicated. Patients with acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL) must be in complete remission at the time of alloHCT(<5% blasts in the bone marrow, normal maturation of all cellular components in the bone marrow and absence of extramedullary disease).
3. Myeloablative conditioning (MAC) regimen, based on Center for International Blood and Marrow Transplant Research (CIBMTR) criteria.
4. T cell-replete peripheral blood graft.
5. Patients must have a matched related or unrelated donor (at least 6/6 match at human leukocyte antigens (HLA) -A, -B and -C for related donors and at least 8/8 match at HLA-A, -B, -C and -DRB1 for unrelated donors).
6. Cardiac function: Left ventricular ejection fraction ≥45% for myeloablative conditioning.
7. Estimated creatinine clearance ≥40 mL/minute (using the Cockcroft-Gault formula and actual body weight).
8. Pulmonary function: Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% (adjusted for hemoglobin) and Forced Expiratory Volume (FEV1) ≥50%.
9. Liver function: total bilirubin <3 x upper limit of normal and alanine aminotransferase (ALT) / aspartate aminotransferase (AST) <5 x upper normal limit.
10. Signed informed consent: Voluntary written consent must be given before patient registration and performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Female patient: A negative pregnancy test will be required for women of child bearing potential. Breast-feeding or lactation is not permitted.
12. Planned posttransplant maintenance therapy is allowed.

Exclusion Criteria:

1. Prior allogeneic HCT.
2. Active central nervous system (CNS) involvement with malignancy.
3. Patients receiving cord blood or haploidentical allograft.
4. Patients undergoing in vivo or ex vivo T cell-depleted alloHCT.
5. Karnofsky Performance Score <60%.
6. Patients with uncontrolled bacterial, viral or fungal infections (currently on treatment and with progression of infectious disease or no clinical improvement) at time of enrollment.
7. Active hepatitis B or C virus infection or known human immunodeficiency virus (HIV) positive.
8. Prior intolerance or allergy to tocilizumab.
9. Use of rituximab, alemtuzumab, anti-thymocyte globulin (ATG) or other monoclonal antibody planned as part of conditioning regimen for GVHD prophylaxis.
10. History of diverticulitis, Crohn's disease or ulcerative colitis.
11. History of demyelinating disorder.
12. Any current uncontrolled cardiovascular conditions, including uncontrolled ventricular arrhythmias, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled angina, or electrocardiographic evidence of active ischemia or active conduction system abnormalities.
13. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R Drobyski, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chhabra S, Szabo A, Clurman A, McShane K, Waters N, Eastwood D, Samanas L, Fei T, Armijo G, Abedin S, Longo W, Hari P, Hamadani M, Shah NN, Runaas L, Jerkins JH, Van den Brink M, Peled JU, Drobyski WR. Mitigation of gastrointestinal graft-versus-host disease with tocilizumab prophylaxis is accompanied by preservation of microbial diversity and attenuation of enterococcal domination. Haematologica. 2023 Jan 1;108(1):250-256. doi: 10.3324/haematol.2022.281309. No abstract available. PMID 36106394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one subjects signed consent, but two did not meet final eligibility criteria and were not enrolled.
Groups:
- Tacrolimus/Methotrexate/Tocilizumab: Patients enrolled on the clinical trial will receive tacrolimus initiating at Day -1 at doses to maintain therapeutic levels per institutional preference and continued until at least Day +90 post-transplant.
  Methotrexate will be administered intravenously and dosed at 15 mg/m2 Day +1 and 10 mg/m2 Days +3, +6 and +11.
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg on Day -1 and at day +100 (+/- 14 days).
  Tacrolimus: Tacrolimus will be given intravenously at a dose of 0.03 mg/kg/day starting Day -3. Subsequent dosing will be based on blood levels.
  Methotrexate: Methotrexate will be administered at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic cell infusion.
  Tocilizumab: Tocilizumab will be administered intravenously (IV) at a dose of 8 mg/kg (maximum dose of 800 mg) once on the Day -1 approximately 24 hours prior to the estimated time of the hematopoietic cell infusion, and subsequently, on Day +100 (+/- 14 days, i.e., Days +86 to +114) post-allogeneic hematopoietic cell transplantation. The infusion will be administered over 60 minutes through a dedicated IV line and must not be administered by IV bolus.
Period: Overall Study
Arm/Group | Tacrolimus/Methotrexate/Tocilizumab
Started | 29
Completed | 26
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus/Methotrexate/Tocilizumab
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With GVHD/Relapse-free (GRFS) Survival
Description: GRFS is defined as survival without grade III-IV acute graft versus host disease (GVHD), systemic therapy requiring chronic GVHD, relapse, or death at 12 months after matched related/unrelated donor bone marrow or peripheral blood allogeneic hematopoietic cell transplantation (alloHCT) using myeloablative conditioning (MAC). Patients who are alive without GVHD will be censored at the last follow-up.
Time Frame: Day 365
Measure: Count of Participants; unit: Participants
Groups:
- Tacrolimus/Methotrexate/Tocilizumab: Patients enrolled on the clinical trial will receive tacrolimus initiating at Day -1 at doses to maintain therapeutic levels per institutional preference and continued until at least Day +90 post-transplant.
  Methotrexate will be administered intravenously and dosed at 15 mg/m2 Day +1 and 10 mg/m2 Days +3, +6 and +11.
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg on Day -1 and at day +100 (+/- 14 days).
  Tacrolimus: Tacrolimus will be given intravenously at a dose of 0.03 mg/kg/day starting Day -3. Subsequent dosing will be based on blood levels.
  Methotrexate: Methotrexate will be administered at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic cell infusion.
  Tocilizumab: Tocilizumab will be administered intravenously (IV) at a dose of 8 mg/kg (maximum dose of 800 mg) once on the Day -1 approximately 24 hours prior to the estimated time of the hematopoietic cell infusion, and subsequently, on Day +100 (+/- 14 days, i.e., Days +86 to +114) post-alloHCT. The infusion will be administered over 60 minutes through a dedicated IV line and must not be administered by IV bolus.
Arm/Group | Tacrolimus/Methotrexate/Tocilizumab
Number analyzed (Participants) | 29
Participants | 25

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tacrolimus/Methotrexate/Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 28/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus/Methotrexate/Tocilizumab (N=29)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Pericardial Tamponade (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Fungal pneumonia
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoman (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus/Methotrexate/Tocilizumab (N=29)
Anemia (Blood and lymphatic system disorders) | 12 (15)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Leukocytosis, <100,000/mm^3
Dry eye (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 8 (9)
Rectal pain (Gastrointestinal disorders) | 2 (3)
Edema limbs (General disorders) | 2 (3)
General disorders - Other, specify (General disorders) | 1 (1) — Subdural Hematoma
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — ENTEROCOLITIS INFECTIOUS
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Enterococcus bacteremia
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — E. Coli
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Rhinovirus
Skin infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (21)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 12 (16)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (8)
Neutrophil count decreased (Investigations) | 21 (61)
Platelet count decreased (Investigations) | 26 (91)
White blood cell decreased (Investigations) | 22 (58)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - Other, pecify (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized muscle weakness
Headache (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT03699631/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT03699631/ICF_001.pdf